CLINICAL TRIAL: NCT05432583
Title: Phase I, Randomized, Observer-blinded, 3-part, Dose Escalation and Expanded Safety and Dose Evaluation Trial to Evaluate the Safety, Tolerability, and Immunogenicity of an Investigational Prophylactic Vaccine for the Prevention of Genital Lesions Caused by Herpes Simplex Virus (HSV)-2 and Potentially HSV-1
Brief Title: A Clinical Trial in Healthy Volunteers and Volunteers With Recurrent Genital Herpes to Study the Safety, Tolerability, and Immune Responses After Vaccination With an Investigational Vaccine Designed to Prevent Genital Herpes Lesions
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: BNT163-01
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Genital Herpes Simplex Type 2
Keywords: Prevention of genital lesions caused by herpes simplex virus-2; Prevention of genital lesions caused by herpes simplex virus-1; Genital infection caused by HSV; Recurrent herpes simplex virus-2 genital herpes; RNA Vaccine; Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: observer-blinded trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A - BNT163 (Experimental): Escalating dose levels
  Interventions: Biological: BNT163
- Part A - Placebo (Placebo Comparator): Isotonic NaCl solution (0.9%)
  Interventions: Other: Placebo
- Part B - BNT163 Dose 1 (Experimental)
  Interventions: Biological: BNT163
- Part B - BNT163 Dose 2 (Experimental)
  Interventions: Biological: BNT163
- Part C - BNT163 (Experimental): One fix dose level of BNT163
  Interventions: Biological: BNT163
- Part C - Placebo (Placebo Comparator): Isotonic NaCl solution (0.9%)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: BNT163 — Anti-viral ribonucleic acid (RNA) vaccine for active immunization against HSV-2 administered as intramuscular injection
  Arms: Part A - BNT163; Part B - BNT163 Dose 1; Part B - BNT163 Dose 2; Part C - BNT163
Other: Placebo — Placebo
  Arms: Part A - Placebo; Part C - Placebo

SUMMARY:
This exploratory trial will have three parts. Part A is a dose escalation part, Part B is an expanded safety and dose evaluation part, and Part C is a safety and immunogenicity evaluation part in individuals with recurrent HSV-2 genital herpes.

Part A will focus on the safety evaluations, and in addition, vaccine-induced immune responses (specifically neutralizing antibodies) will also be analyzed to assess if there is a dose-response.

Part B of the trial will expand the safety characterization for two dose levels of BNT163 selected based on Part A data and will also enable a more comprehensive assessment of the impact of pre-existing immunity to HSV-1 and -2 on the safety and immune responses to BNT163.

Part C will evaluate safety and immunogenicity of BNT163 compared to a placebo in a three-dose regimen in participants with a history of HSV-2 recurrent genital herpes.

DETAILED DESCRIPTION:
In Part A, participants will be randomized 5:1 to BNT163:placebo. In Part B, participants will be randomized 1:1 to either of the two selected dose levels based on data from Part A. In Part C, participants will be randomized 1:1 to BNT163:placebo.

In Part A & B, participants will receive three intramuscular doses of a fixed dose level of the BNT163 vaccine (Part A and B) or placebo (Part A only).

In Part C, participants will receive three intramuscular doses of one fixed dose level of the BNT163 vaccine or placebo. In this part, continuous suppressive antiviral therapy is given over the entire vaccine dosing period (during and between vaccine doses) to prevent administration of the vaccine concomitantly to viral replication and active genital herpes.

ELIGIBILITY:
Inclusion Criteria (applicable to all participants and all parts unless otherwise specified):

* Have given informed consent by signing and dating the informed consent form (ICF) before initiation of any trial-specific procedures.
* Are aged 18 to 55 years, have a body mass index over 18.5 kg/m^2 and under 35 kg/m^2 and weigh at least 50 kg at Visit 0.
* Are willing and able to comply with scheduled visits, treatment schedule, laboratory tests, and other requirements of the trial. This includes that they are able to understand and follow trial-related instructions.
* Are overall healthy in the clinical judgment of the investigator based on medical history, physical examination, 12-lead electrocardiogram (ECG), vital signs, and screening laboratory tests (blood clinical laboratory) at Visit 0 (for Part C only: (all results must be available prior to Pre-dose Visit 1).
* Part C only: Have had

  * a diagnosis (>1 year) of genital herpes confirmed in medical records; and
  * with at least 3 and no more than 9 participant-reported genital herpes recurrences either in the 1 year preceding Visit 0, or, if currently on continuous antiviral therapy, in the 1 year preceding the start of continuous antiviral therapy.
* Part C only: Are seropositive for HSV-2 as determined by Western Blot (result must be available prior to Pre-Dose Visit 2).
* Part C only: Are willing to comply with the protocol-specified schedule for continuous antiviral therapy.
* Part C only: Are willing to refrain from the use of episodic antiviral therapy according to the antiviral therapy schedule. Episodic antiviral therapy may be used outside the prohibited periods.
* Negative human immunodeficiency virus (HIV)-1 and HIV-2 blood test at Visit 0.
* Negative Hepatitis B surface antigen at Visit 0.
* Negative anti-Hepatitis C virus (HCV) antibodies (anti-HCV), or undetectable HCV viral load if the anti-HCV is positive at Visit 0.
* Negative syphilis test at Visit 0.
* Volunteers of childbearing potential (VOCBP): negative serum beta human chorionic gonadotropin (β-HCG) pregnancy test at Visit 0 and negative urine pregnancy test prior to each investigational medicinal product (IMP) administration and at the end of the trial. Volunteers born female that are postmenopausal (verified by follicle stimulating hormone [FSH] level) or permanently sterilized (verified by medical records) will not be considered VOBCP.
* VOCBP who agree to practice a highly effective form of contraception and to require their male partners to use condoms coated with a spermicidal agent, starting at Visit 0 and continuously until 60 days after receiving the last trial treatment.
* VOCBP who agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during trial, starting at Visit 0 and continuously until 60 days after receiving the last trial treatment.
* Men who are sexually active with a VOCBP and have not had a vasectomy who agree to use condoms coated with a spermicidal agent and to practice a highly effective form of contraception with their partners of childbearing potential during the trial, starting at Visit 0 and continuously until 90 days after receiving the last trial treatment.
* Men who are willing to refrain from sperm donation, starting at Visit 0 and continuously until 90 days after receiving the last trial treatment.

Exclusion Criteria (applicable to all participants and all parts unless otherwise specified):

* Breastfeeding or intending to become pregnant within the projected duration of the trial starting with Visit 0 until 60 days after receiving the last trial treatment or intending to father children within the projected duration of the trial starting with Visit 0 until 90 days after receiving the last trial treatment.
* Part A & B only: Current or history of symptomatic genital herpes infections. Volunteers with oral herpes or herpetic whitlow will not be excluded.
* Current or history of any form of ocular HSV infection or HSV-related central nervous system disease or complication.
* History of any serious adverse reactions to vaccines or to vaccine components such as lipids, and including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain.
* Current or history of the following medical conditions:

  * Uncontrolled or moderate or severe respiratory diseases (e.g., asthma, chronic obstructive pulmonary disease); symptoms of asthma severity as defined in the most recent National Asthma Education and Prevention Program Expert Panel report;
  * History of thyroidectomy, or thyroid disease requiring medication during the last 12 months;
  * History of diabetes mellitus type 1 or type 2, including cases controlled with diet alone (not excluded: history of isolated gestational diabetes);
  * Hypertension (elevated blood pressure or hypertension during screening or previously that is not well controlled only [consistently ≤140 mm Hg systolic and ≤90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be ≤150 mm Hg systolic and ≤90 mm Hg diastolic at enrollment] or if systolic blood pressure ≥150 mm Hg at enrollment or diastolic blood pressure ≥100 mm Hg confirmed by two measurements prior to enrollment);
  * Malignancy within 5 years of Visit 0, excluding localized basal or squamous cell cancer;
  * Current or history of cardiovascular diseases, e.g., myocardial infarction, congestive heart failure, cardiomyopathy, or clinically significant arrhythmias, myocarditis, or pericarditis;
  * Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions);
  * Seizure disorder: History of seizure(s) within past 3 years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* History of psychiatric illness, including alcohol abuse or drug addiction within 1 year before Visit 0, or a history (within the past 5 years) of substance abuse or known medical, psychological, or social conditions which, in the opinion of the investigator, could compromise their wellbeing if they participate as participants in the trial, or that could prevent, limit, or confound the protocol specified assessments.
* Any of the following associated with immune dysregulation:

  * Primary immunodeficiencies.
  * History of solid organ or bone marrow transplantation.
  * Asplenia: any condition resulting in the absence of a functional spleen.
  * Currently existing or history of autoimmune disease including and not limited to thyroid autoimmune disease, multiple sclerosis, psoriasis, etc.
* Use of any non-trial IMP within 28 days before Dose 1 (Visit 1) (Parts A & B) or before Pre-dose Visit 2 (Part C) in this trial or planned receipt continuously until Visit 6 (Part C) or Visit 12 (Parts A & B) in this trial, or participation in the active treatment phase of another interventional clinical trial.
* Previous vaccination with an investigational herpes virus vaccine at any time.
* Any non-trial vaccination with a licensed live attenuated vaccine within 28 days before and after each dose, or within 14 days before and after each dose for all other licensed vaccines.
* Received allergy treatment with antigen injections within 28 days before first IMP administration or that are scheduled within 14 days after Visit 1.
* Received blood/plasma products or immunoglobulin within 120 days before Visit 1 or planned administration starting at Visit 0 until completion of Visit 6 (Part C) or Visit 12 (Parts A & B).
* Part A & B only: Received chronic suppressive antiviral therapy for treatment of recurrent HSV-1 and/or HSV-2 genital herpes infections (i.e., oral acyclovir, oral valacyclovir, oral famciclovir, and/or intravenous ganciclovir) from 1 year prior to Visit 0 until completion of Visit 12.
* Any existing condition which may affect vaccine injection and/or assessment of local reactions assessment at the injection site, e.g., tattoos, severe scars.
* Vulnerable individuals as per International Council for Harmonisation (of Technical Requirements for Pharmaceuticals for Human Use) (ICH) E6 definition, i.e., are individuals whose willingness to volunteer in a clinical trial may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate. This includes investigator site staff directly involved in the conduct of the trial and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the trial and their family members.
* Part A & B only: Any screening hematology and/or blood chemistry laboratory value that meets the definition of a Grade ≥2 abnormality at Visit 0. For laboratory values for which toxicity grading guidance is not available or for Grade ≤1 abnormalities, participant eligibility will be determined at the discretion of the investigator.
* Part C only: Any screening hematology and/or blood chemistry laboratory value that meets the definition of a Grade ≥3 abnormality at Visit 0. Grade 2 abnormal laboratory values may be retested; if the result is confirmed, the participant must be excluded. For laboratory values for which toxicity grading guidance is not available, or for Grade ≤1 abnormalities, participant eligibility will be determined at the discretion of the investigator.
* Part B only: Applicable HSV serology stratum is already full or the HSV serostatus is reported as indeterminate.
* Part C only: At the end of the first 28-day swabbing period, a participant has submitted fewer than 45 swabs.
* Part C only: If a participant has evidence of active genital herpes infection (prodrome or lesions) at the Dose 1 visit which had already been delayed due to presence of lesions at previously scheduled Dose 1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 318 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Frequency of solicited local reactions at the injection site (pain, erythema/redness, induration/swelling) recorded up to 7 days after each dose | Up to 7 days after each dose
  For each dose level (DL) per BNT163 dosing schedule and for the combined placebo group.
Frequency of solicited systemic reactions (vomiting, diarrhea, headache, fatigue/tiredness, myalgia, arthralgia, chills, and fever) recorded up to 7 days after each dose | Up to 7 days after each dose
  For each DL per BNT163 dosing schedule and for the combined placebo group.
Percentage of participants with at least one unsolicited adverse event (AE) occurring up to 28 days after each dose | From Day 1 up to Day 197
  For each DL per BNT163 dosing schedule and for the combined placebo group.
Percentage of participants in each cohort with at least one serious AE, or AE of special interest, or medically attended AE occurring up to 24 weeks post-Dose 3 (Parts A & B) or post-Dose 2 (Part C) | From Day 1 up to Day 337
  For each DL per BNT163 dosing schedule and for the combined placebo group.
Number of unsolicited AEs occurring up to 28 days after each dose | From Day 1 up to Day 197
  For each DL per BNT163 dosing schedule and for the combined placebo group.
Percentage of unsolicited AEs occurring up to 28 days after each dose | From Day 1 up to Day 197
  For each DL per BNT163 dosing schedule and for the combined placebo group.

SECONDARY OUTCOMES:
Geometric mean titer (GMT) at each time point | From Day 1 up to Day 337
  HSV-2 glycoproteins (g)C2, gD2, and gE2 binding antibody titers enzyme-linked immunosorbent assay (ELISA). HSV-2 neutralizing antibody titers.
  For each DL per BNT163 dosing schedule at baseline, 7 days (Parts A & B only) and 28 days after each dose and at 24 weeks post-Dose 3 (all parts) and for the combined placebo group.
Geometric mean fold (GMF) change from baseline of neutralizing and binding antibody titers to each time point after vaccination | From Day 1 up to Day 337
  HSV-2 gC2, gD2, and gE2 binding antibody titers ELISA. HSV-2 neutralizing antibody titers.
  For each DL per BNT163 dosing schedule at baseline, 7 days (Parts A & B only) and 28 days after each dose and at 24 weeks post-Dose 3 (all parts) and for the combined placebo group.
Part A and B only - Percentage of participants with seroconversion defined as a minimum of 4-fold increase from baseline of neutralizing and binding antibody titers to each subsequent time point after vaccination | From Day 1 up to Day 337
  For each DL per BNT163 dosing schedule at baseline, 7 days (Parts A & B only) and 28 days after each dose and at 24 weeks post-Dose 3 (all parts) and for the combined placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (6):
- United States (6):
  - Alliance for Multispecialty Research, LLC, Tempe, Arizona
  - Great Lakes Clinical Trials - Flourish Research, Chicago, Illinois
  - Accellacare Raleigh Medical Group, Raleigh, North Carolina
  - Accellacare PMG Research Wilmington LLC, Wilmington, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No